CLINICAL TRIAL: NCT01416610
Title: A Prospective, Observational, Multicenter Non-interventional Trial Examining Efficacy of Combination Therapy With PEGASYS® (Peginterferon Alfa-2a 40KD) Plus COPEGUS® (Ribavirin) in Patients With Chronic Hepatitis C, Genotype 2, 3, 1 or 4, Undergoing an Opioid Maintenance-Therapy With Special Focus on Patient Compliance and Quality of Life
Brief Title: An Observational Study of Pegasys (Peginterferon Alfa-2a) Plus Copegus (Ribavirin) in Participants With Chronic Hepatitis C (CHC), Genotype 2, 3, 1 or 4, Undergoing Opioid Maintenance Therapy
Acronym: PEGHOPE
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25159
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Participants with chronic hepatitis C, Genotype 2, 3, 1 or 4, undergoing an opioid maintenance therapy

SUMMARY:
This prospective, multi-center, observational study will evaluate the efficacy and safety of Pegasys (peginterferon alfa-2a) plus Copegus (ribavirin) in participants with previously untreated chronic hepatitis C, genotype 2, 3, 1 or 4, who are undergoing opioid maintenance therapy. Data will be collected from eligible participants receiving Pegasys and Copegus treatment as prescribed by treating physician and treatment-free follow-up period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Participants undergoing an opioid maintenance therapy
* Serologic evidence of CHC prior to therapy
* CHC genotype 2, 3, 1 or 4
* Quantifiable serum hepatitis C (HCV) ribonucleic acid (RNA)
* All fertile males and females receiving ribavirin must use two forms of effective contraception during treatment with study drugs and for 7 months after completion of treatment

Exclusion Criteria:

* Harmful use of psychoactive substances (including excessive alcohol consumption) that precludes successful participation in the study at the discretion of the investigator
* Pegylated interferon, standard interferon or ribavirin therapy at any time prior to initiation of the study
* Co-infection with hepatitis A, hepatitis B or Human Immunodeficiency Virus (HIV)
* Current diagnosis of a major depression or any psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic hepatitis C (CHC), Genotype 2, 3, 1 or 4, undergoing an opioid maintenance therapy
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2010-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Austria (10):
  - Lkh Hoergas-Enzenbach; Abt. Für Innere Medizin, Gratwein
  - Lkh-Univ. Klinikum Graz, Graz
  - Lkh innsbruck - univ. Klinikum innsbruck - Tiroler landeskrankenanstalten ges.m.b.h.; Innere Medizin, Innsbruck
  - Klinikum Klagenfurt am Wörthersee; 2. Medizinische Abteilung, Klagenfurt
  - A.Ö. Krankenhaus Der Elisabethinen Linz; Iv. Med. Abtl., Linz
  - Gesundheitszentrum Wien Mitte, Vienna
  - Krankenanstalt Rudolfstiftung; Iv. Med. Abtl., Vienna
  - Medizinische Universität Wien; Univ.Klinik für Innere Medizin III - Gastroenterologie & Hepatologie, Vienna
  - Kaiser Franz Josef Spital; Iv. Medizinische Abt., Vienna
  - Wilhelminenspital; 6. Medizinische Abteilung Wilhelminenspital; 6. Medizinische Abteilung, Vienna

REFERENCES:
- [Derived] Gschwantler M, Laferl H, Vogel W, Korak W, Moser S, Hofer H, Bauer B, Schleicher M, Bognar B, Bischof M, Stauber R, Maieron A, Ferenci P; Austrian Hepatitis Study Group. Efficacy of peginterferon plus ribavirin in patients receiving opioid substitution therapy : Final results of the Austrian PegHope study. Wien Klin Wochenschr. 2018 Jan;130(1-2):54-61. doi: 10.1007/s00508-017-1263-2. Epub 2017 Sep 12. PMID 28900714

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 88
Intention to Treat | 88
Safety Population | 86
Per Protocol | 83
Completed Treatment | 47
Completed Follow-up | 45
Completed | 45
Not Completed | 43
Not completed — Adverse Event | 4
Not completed — Adverse Event -Patient decision | 3
Not completed — Lack of Efficacy | 4
Not completed — No reason given | 5
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 7
Not completed — Sufficient treatment duration (PCR neg.) | 7

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 64
Region of Enrollment [Number; unit: participants]
  Austria | 88

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response 24 Weeks After Completing Treatment (SVR24)
Description: SVR24 is defined as percentage of participants with undetectable Hepatitis C virus (HCV) ribonucleic acid (RNA) 24 weeks after completing treatment, using a last observation carried forward (LOCF) approach. Percentage is based on the number of non-missing observations (total).
Time Frame: 24 weeks after completing treatment, within 3 years, 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 88
percentage of participants | 83.0 [73.8 to 89.4]

2. Secondary Outcome: Percentage of Participants With SVR 12
Description: SVR 12 is defined as percentage of participants with undetectable HCV RNA 12 weeks after completing treatment, using a LOCF approach. Percentage is based on the number of non-missing observations (total).
Time Frame: 12 weeks after completing treatment, within 3 years, 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 88
percentage of participants | 81.8 [72.5 to 88.5]

3. Secondary Outcome: Percentage of Participants With End of Treatment Response
Description: A participant was considered to have end of treatment response if there was undetectable HCV RNA after completing treatment, using a LOCF approach. Percentage is based on the number of non-missing observations (total).
Time Frame: at end of treatment, within 3 years, 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 88
percentage of participants | 87.5 [79.0 to 92.9]

4. Secondary Outcome: Percentage of Participants With Virological Relapse
Description: Virological relapse is defined as no SVR24 in a participant with undetectable HCV RNA at end of treatment who has at least one post-treatment polymerase chain reaction (PCR) result available, using a LOCF approach. Percentage is based on the number of non-missing observations (total).
Time Frame: by end of follow-up, within 3 years, 6 months
Population: Participants who completed treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 47
percentage of participants | 10.6 [4.6 to 22.6]

5. Secondary Outcome: Short Form Health Survey (SF-36) Scores by Visit
Description: The SF-36 questionnaire items were scored and transformed according to the SF-36 Health Survey Manual & Interpretation Guide. Summary scores for SF-36 dimensions of physical functioning, role functioning, bodily pain, general health, vitality, social functioning, and mental health were scored on a scale of 0 (worst) to 100 (best), and health transition was scored on a scale of 0 (worst) to 5 (best). Summary SF-36 scores are reported by category and by visit.
Time Frame: at baseline, week 12, end of treatment and end of follow-up within 3 years, 6 months
Population: Participants with a viable score at the given time point
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline: Baseline Visit
- Week 12: Week 12 Visit
- End of Treatment: End of Treatment Visit
- End of Follow-up: End of Follow-up Visit
Arm/Group | Baseline | Week 12 | End of Treatment | End of Follow-up
Number analyzed (Participants) | 88 | 88 | 88 | 88
units on a scale
  Physical Functioning (n=54,34,37,22) | 77.9 (21.7) | 63.5 (25.1) | 62.7 (22.3) | 76.1 (26.5)
  Role Functioning - Physical (n=52,34,37,22) | 60.6 (40.9) | 32.4 (37.7) | 24.3 (37.0) | 70.5 (39.1)
  Bodily Pain (n=53,35,37,22) | 70.8 (27.7) | 58.7 (29.3) | 52.5 (27.8) | 75.4 (29.7)
  General Health (n=50,35,36,22) | 50.9 (18.9) | 46.1 (18.6) | 50.5 (18.7) | 65.4 (19.3)
  Vitality (n=52,35,37,22) | 42.8 (21.5) | 26.1 (19.3) | 33.9 (20.2) | 48.6 (20.0)
  Social Functioning (n=53,35,37,23) | 69.8 (27.1) | 52.5 (28.6) | 48.0 (27.4) | 72.3 (32.6)
  Role Functioning - Emotional (n=53,34,36,22) | 57.2 (44.0) | 31.4 (37.6) | 31.5 (36.5) | 69.7 (37.0)
  Mental Health (n=52,34,37,22) | 59.1 (19.2) | 49.4 (19.8) | 51.7 (22.4) | 67.2 (25.7)
  Reported Health Transition (n=54,34,37,22) | 3.3 (1.2) | 3.6 (1.2) | 3.2 (1.5) | 2.0 (1.2)

6. Secondary Outcome: Fatigue Severity Scale (FSS) Score by Visit
Description: The Fatigue Severity Scale (FSS) consists of 9 questions, each answered within a range of 1-7, where lower scores indicate less fatigue in everyday life. The FSS score is the mean of the 9 numbers. Mean scores are presented by visit.
Time Frame: at baseline, week 12, end of treatment and end of follow-up within 3 years, 6 months
Population: Participants with a viable score at the given time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 88
units on a scale
  Baseline (n=56) | 4.0 (1.4)
  Week 12 (n=35) | 5.0 (1.3)
  End of treatment (n=37) | 5.0 (1.4)
  End of follow-up (n=24) | 3.8 (1.8)

7. Secondary Outcome: Beschwerdeliste (BL) Score by Visit
Description: The BL questionnaire items were scored by calculating the average response to all answered items. Items can be graded 1="stark" (affliction is strong) to 4="gar nicht" (not present). The higher the BL score, the less afflictions were present for a participant. Mean scores are presented by visit.
Time Frame: at baseline, week 12, end of treatment and end of follow-up within 3 years, 6 months
Population: Participants with a viable score at the given time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 88
units on a scale
  Baseline (n=59) | 3.1 (0.5)
  Week 12 (n=34) | 2.8 (0.5)
  End of treatment (n=36) | 2.7 (0.5)
  End of follow-up (n=24) | 3.1 (0.6)

8. Secondary Outcome: Beck Depression Inventory (BDI) Score by Visit
Description: The BDI questionnaire items were scored by generating the sum of the responses to all answered items. Each result was categorized into one of four categories: 0-13= no depression or clinically not significant or in remission; 14-19= mild depression; 20-28= moderate depression; or 29-63= severe depression. Mean scores are presented by visit.
Time Frame: at baseline, week 12, end of treatment and end of follow-up within 3 years, 6 months
Population: Participants with a viable score at the given time point
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 88
units on a scale
  Baseline (n=50) | 13.7 (9.0)
  Week 12 (n=33) | 18.4 (11.1)
  End of treatment (n=33) | 16.9 (9.4)
  End of follow-up (n=22) | 11.6 (10.7)

ADVERSE EVENTS:
Groups:
- Safety Population: Participants who started treatment
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 14/86
Other Adverse Events (participants affected / at risk) | 60/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=86)
Abscess limb (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Drug withdrawal syndrome (General disorders) | 2
Anorexia nervosa (Psychiatric disorders) | 1
Withdrawal syndrome (Psychiatric disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Uterine cyst (Reproductive system and breast disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=86)
Fatigue (General disorders) | 42
Influenza like illness (General disorders) | 14
Pyrexia (General disorders) | 10
Depression (Psychiatric disorders) | 23
Insomnia (Psychiatric disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 15
Decreased appetite (Metabolism and nutrition disorders) | 15
Headache (Nervous system disorders) | 14
Nausea (Gastrointestinal disorders) | 13
Weight decreased (Investigations) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.